CLINICAL TRIAL: NCT00822822
Title: Evaluation of Patient Functionality and Utility of Web-Based Personal Health History and Risk Assessment
Brief Title: Evaluation of Patient Functionality and Utility of Web-Based Personal Health History and Risk Assess
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-14731; 104330 (Other: USF IRB)
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2010-10

CONDITIONS: Cancer; Cancer Screening Patients; Patient Volunteers
Keywords: Questionnaire; Electronic Health History
MeSH Terms: conditions — Neoplasms | interventions — Health Records, Personal

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Health History Process
  Interventions: Behavioral: First Questionnaire; Behavioral: Health History; Behavioral: Second Questionnaire

INTERVENTIONS:
Behavioral: First Questionnaire — Complete questionnaire before completing health history
Behavioral: Health History — Complete electronic health history
Behavioral: Second Questionnaire — Complete questionnaire after completing electronic health history

SUMMARY:
The purpose of this research study is to find out what Moffitt and Lifetime patients think of the electronic medical records process.

DETAILED DESCRIPTION:
Patient will complete a questionnaire about their knowledge of computers and how long they think it will take them to finish the patient health history using a computer.

Patient will complete the electronic record carefully and tell us if they had any difficulties, questions or comments about the format.

Patient will answer a questionnaire about how well they liked or did not like using the electronic system to give their health history.

Participation in this study will take approximately 30 minutes to 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* The breakdown of patients recruited by stratified dimensional sampling. Overall, we will attempt to equally recruit patients from the unique strata for each domain evaluation in this study. Patients health status will be determined by the ECOG Performance status . We assume that all patients being seen at the Lifetime Cancer Screening and Prevention center will be of good to fair health, while patients seen at the Cancer hospital will range from good- to- fair to poor health status. Gender is also used as a sampling factor because there are modules within this web-based health history forms that are specific for each gender.

Exclusion Criteria:

* Respondents who refuse to participate or who become too ill at any point in the assessment, will be excluded. Non-English speaking patients will be excluded. Names and other identifying information will not be collected and all data will be reported in aggregate form. Due to the nature of our stratified samples strategy, some patients will be excluded if they meet the criteria for a recruitment stata, but that stata is full.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People receiving services at Moffitt Cancer Center or Lifetime Cancer Screening Center
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2006-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Create a system for collecting patient health histories that may be beneficial to patients and people receiving services at Moffitt Cancer Center or Lifetime Cancer Screening Center | 1 hour per participant

CONTACTS AND LOCATIONS:
Overall Officials: Erin Siegel, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States